CLINICAL TRIAL: NCT05308589
Title: Continuous Postoperative Pericardial Flushing After General Cardiac Surgery Procedures With the Haermonics Investigational Device: Study Protocol of the FLUID (FLUsh With Investigational Device) Trial
Brief Title: CPPF After General Cardiac Surgery
Acronym: FLUID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study no longer fits our strategic goals. The preliminary results of FLUID have led to an improved version of the current device. We believe it is necessary to initiate a new study, with the improved version of the device.
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Haermonics BV (Industry); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Eva Diephuis, Medical doctor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL74428
Record Dates: First submitted 2022-02-28; First posted 2022-04-04 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Surgical Procedures; Retained Blood Syndrome; Cardiac Tamponade; Postoperative Hemorrhage
Keywords: Continuous Postoperative Pericardial Flush (CPPF); CABG; Retained Blood Syndrome; Chest tubes [Mesh]; Blood Transfusion [mesh]; Therapeutic irrigation [Mesh]
MeSH Terms: conditions — Cardiac Tamponade; Postoperative Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Postoperative Pericardial Flushing (Experimental): Continuous Postoperative Pericardial Flushing (inflow of 500 ml NaCl 0,9% flushing fluid into the pericardial cavity during the first 8 postoperative hours) executed with the Haermonics investigational device
  Interventions: Device: CPPF
- Control (No Intervention): Standard care

INTERVENTIONS:
Device: CPPF — Continuous Postoperative Pericardial Flush
  Arms: Continuous Postoperative Pericardial Flushing

SUMMARY:
In two randomized clinical trials the investigators have demonstrated that continuous postoperative pericardial flushing (CPPF) therapy can reduce postoperative blood loss and bleeding-related complications after cardiac surgery and that CPPF therapy is safe and feasible in an experimental setting. The Haermonics investigational device is a novel medical device that enables CPPF therapy to be used in daily clinical setting. The aim of this study is three-fold. First, to evaluate the safety and functionality of the Haermonics investigational device. Secondly, to investigate the effect of CPPF therapy on bleeding related complications in the adulty cardiac surgery population. Thirdly, to explore the effect of CPPF therapy on intraluminal chest tube clogging.

DETAILED DESCRIPTION:
CPPF therapy

Prolonged or excessive bleeding after cardiac surgery can lead to a broad spectrum of secondary complications. One of the underlying causes is incomplete wound drainage, with subsequent accumulation of blood and clots in the pericardium. It has been demonstrated that this retained blood and clots lead to even more fibrinolytic activity in the mediastinum and pericardial space, and therefore may contribute to increased or prolonged bleeding. Based on this principle, the method of continuous postoperative pericardial flushing (CPPF) has been invented and further developed. The hypothesis is that CPPF therapy works by mechanical cleaning properties and by diminishing fibrinolysis and inflammation. The CPPF protocol includes the inflow of NaCl 0,9% flushing fluid into the pericardial cavity during the first postoperative hours in patients who underwent cardiac surgery. In this way, the blood and clot mixture can be diluted into a lower viscosity solution, thereby enhancing the evacuation of blood and clots from the pericardial space and preventing chest tube obstruction.

The Haermonics investigational device

Because CPPF therapy includes the dilution of the normal postoperative mediastinal chest tube drainage (MCTD), the clinical assessment of the exact amount of blood loss is more difficult. Yet, blood loss is an important factor in clinical decision making, namely the decision if the patient needs a surgical re-exploration for postoperative bleeding or not. Roughly, in patients who receive CPPF therapy, blood loss can be estimated by extracting the total inflow flushing volume from the total MCTD. This method was used in the experimental setting of the previous CPPF trails but is considered unsuitable for use in daily practice because of three reasons. First, the required registration of in- and outflow volume is labour intensive. Secondly, because this registration can only be done intermittently, which can be dangerous in case of a fast bleeding rate. Thirdly, blood loss calculation could potentially be inaccurate because sometimes, clinically insignificant, amounts of flushing fluid are retained or absorbed in the pericardial or pleural spaces, thereby making the blood loss calculation inaccurate.

The first commercial Haermonics device will have four essential functionalities that make CPPF therapy safe and feasible for daily clinical use. 1) Automatic monitoring of the outflow volume, 2) Quantification of the content of the outflow volume by means of real time and continuous haematocrit (hct) analysis of the MCTD, 3) Warming of the flushing fluid to body temperature and temperature measurements of the flushing fluid, and 4) Continuous intrapericardial pressure measurement. The investigational device that will be used in this study will have all these functionalities, but available data will not be used for clinical decision making yet.

Previous studies

CPPF, executed with a researcher instead of a medical device, has been investigated in two randomized clinical trials. The CPPF protocol included the inflow of 500 ml NaCl 0,9% flushing fluid into the pericardial cavity during the first 12 postoperative hours in patients who underwent cardiac surgery. In this way, the blood and clot mixture were diluted into a lower viscosity solution, thereby enhancing the evacuation of blood and clots from the pericardial space and preventing chest tube obstruction. In two distinct cardiac surgery populations, both trials showed CPPF led to a statistically significant reduction in the primary outcome, i.e., blood loss, while pooled data showed a statistically significant difference for the clinically most relevant secondary end points, like the incidence of re-interventions for either non-surgical bleeding and/or acute cardiac tamponade (0 vs. 8 in CPPF vs. control group).

The present study is powered to assess the effects of CPPF, executed by the Haermonics investigational device, in comparison with standard care on these clinically more relevant endpoints in a population of adult cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject should be scheduled for a general cardiothoracic surgery procedure with the use of cardiopulmonary bypass, amongst others, the main categories are;

* Coronary artery bypass grafting (CABG),
* Valve surgery,
* CABG combined with valve surgery
* Elective patients scheduled for aortic surgery (including valve sparing root replacement (VSRR), Bentall procedures, ascending aorta- aortic arch replacement)

Including the initial study population:

* Patients scheduled for CABG with continued DAPT
* Patients with aIE scheduled for valve replacement
* Patients scheduled for complex or multiple cardiac (redo) procedures with an (expected) CPB time >300 minutes
* Patients undergoing aortic surgery with DHCA

Exclusion Criteria:

* Euroscore II > 20%
* Intraoperatively diaphragm injury leading to an open connection between the thoracic and abdominal cavity
* Age < 18
* Inability to understand study information
* Participation in any study involving an investigational drug or device
* Emergent procedures
* Procedures performed off pump, without the use of cardiopulmonary bypass.
* Minimal invasive cardiac surgery procedures (e.g. minithoracotomy and hemisternotomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Incidence of re-exploration | 7 days
  The incidence of re-exploration for either cardiac tamponade and/or excessive bleeding due to non-surgical bleeding.

SECONDARY OUTCOMES:
To assess safety and feasibility of the Haermonics investigational device | 8 hours
  Incidence of treatment related serious Adverse Events
Hct-sensor validation | 8 hours
  comparibility of the hct values of the chest drain volume measured by the Haermonics investigational device (hourly during the first 10 hours in the ICU and at chest tube removal) and hct values of chest drain samples (drawn from the outflow tube during the first 10 hours in the ICU and at chest tube removal) performed by the local laboratory.
Number of participants with new onset postoperative fibrillation requiring medical therapy or electrocardioversion (ECV) | during hospital stay, average of 3-7 days
  incidence of new onset postoperative fibrillation requiring medical therapy or electrocardioversion (ECV)
To investigate the clinical effects of CPPF on the use of blood products and administration of coagulation factors | during hospital stay, average of 3-7 days
  Number of participants that reveived blood products and/or coagulation factors
To investigate the clinical effects of CPPF on the use of blood products and administration of coagulation factors | during hospital stay, average of 3-7 days
  Number of units per patients
To investigate the clinical effects of CPPF on ICU and hospital stay | during hospital stay, average of 3-7 days
  hospital stay in the operating hospital (days)

OTHER OUTCOMES:
To assess cost-effectiveness | 3 months
  costs per QALY gained using the EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: R. Klautz, Prof, Principal Investigator — Amsterdam UMC
Locations (4):
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Leiden University Medical Center, Leiden
  - St. Antonius Ziekenhuis, Nieuwegein